CLINICAL TRIAL: NCT07114445
Title: The Effect of Diabetic Foot Training Given to Patients With Type-2 Diabetes Using Virtual Reality Glasses on Foot Care Behaviors
Acronym: Diabetes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, SEDA ILGUN, PhD student, principal investigator, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GAZİANTEP U
Record Dates: First submitted 2025-05-28; First posted 2025-08-11 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Prevention of Diabetic Foot
Keywords: virtual reality, diabetic foot training

STUDY DESIGN:
Intervention Model Description: Before the study, patients will be informed and their consent will be obtained. After dividing the patients into intervention and control groups, the researcher will administer data collection forms (questionnaire and Foot Care Behavior Scale (FBS) to both groups before the training. Patients in the intervention group will receive preventive diabetic foot training using virtual reality goggles. Patients in the intervention group will be invited to the hospital at baseline, 4th, 8th, 12th, and 24th weeks. Training will be repeated using virtual reality goggles each week, after which the FBS (Foot Care Behavior Scale) will be administered. The 5-point Likert-type scale adapted for the Foot Care Behavior Scale (FBS) consists of a single dimension and 15 items (1= Never, 2= Occasionally, 3= Sometimes, 4= Often, and 5= Always). The lowest possible score on the scale is 15, and the highest is 75. Higher scale scores indicate better foot self-care behaviors.
Masking Description: No application will be made other than the routine treatment and care of the clinic, and questionnaires will be applied simultaneously with the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Glasses Education Group (Experimental): Patients in the intervention group will be called to the hospital at baseline, weeks 4, 8, 12, and 24 as part of routine checkups based on the educational content developed in line with the literature. The diabetic foot training will be repeated using virtual reality glasses, followed by the foot care behavior scale. Data collection forms will be administered to the patients by the researchers using a face-to-face interview technique, lasting approximately 15-20 minutes.
  Interventions: Other: Diabetes Treatment
- Kontrol grubu (No Intervention): Patients in the control group will not receive any intervention other than the routine practices of the clinic, and data collection tools will be applied when they come to the polyclinic for routine check-ups simultaneously with the intervention group. At the end of the study, patients in the control group will also receive one diabetic foot training with virtual reality glasses.

INTERVENTIONS:
Other: Diabetes Treatment — Training with virtual reality glasses
  Arms: Virtual Glasses Education Group

SUMMARY:
Diabetes mellitus is a chronic disease characterized by high blood sugar resulting from insulin deficiency and/or ineffectiveness. Diabetes is increasingly recognized as a significant public health problem due to its increasing prevalence and potential for a wide range of complications. Diabetic foot, one of the most common complications of diabetes, has become a widespread problem in parallel with the rapidly increasing prevalence of diabetes both globally and domestically. Since healthcare expenditures for diabetic foot care account for one-third of total spending on diabetes treatment, the importance of planning patient education, implementing evidence-based preventive approaches, and regularly monitoring patients to prevent the development of diabetes and diabetic foot is evident. Furthermore, the adoption of evidence-based preventive approaches and regular patient follow-up are essential in this context. Diabetes education nurses, in particular, play a critical role in this regard. Today, with advancements in health technologies and diabetes treatments, significant breakthroughs and improvements in diabetes treatment and care are regularly occurring. Therefore, nurses should plan and implement training every six months or even annually to share current information with patients and facilitate their adaptation to new treatment approaches. The literature particularly emphasizes the importance of providing comprehensive education to individuals with diabetes on disease management, including diet, medication, exercise, and foot care. The need to address the specific needs of these patients for optimal care is also emphasized. Therefore, it is crucial to design and implement effective educational strategies that incorporate current technological applications to transform the knowledge and habits of individuals with diabetes into adaptive behaviors that can reduce the likelihood of developing diabetic foot ulcers. One such application, virtual reality headsets, provide an immersive, three-dimensional virtual environment with high-quality visuals and audio, enabling individuals to learn through experiential learning by simulating realistic scenarios. This application can also increase patients' skill proficiency and motivation. However, our review of the relevant literature revealed no studies using virtual reality headsets as a method for providing diabetic foot education. In light of the above, this study, which examines the impact of diabetic foot education provided to patients via virtual reality headsets on foot care behaviors, is expected to be unique compared to similar studies. The research results are expected to contribute significantly to the prevention of diabetic foot ulcers and the provision of optimum diabetic foot care.

DETAILED DESCRIPTION:
Developing preventive diabetic foot care practices in a virtual environment and demonstrating them to patients using VR headsets: An educational video prepared in a virtual environment based on literature and expert opinions (the educational content was developed in accordance with the Printable Materials Patient Education Material Assessment Tool (HEMDA-B) by consulting an endocrinologist, a podiatrist, a diabetes education nurse, and nine faculty members from various universities). This video will be integrated into VR headsets and demonstrated to patients. The educational content will cover the importance of diabetes and the diabetic foot, risk factors for the diabetic foot, the causes of diabetic foot and diabetic foot symptoms, preventive foot care behaviors, how to perform a self-foot examination, proper nail care, choosing appropriate socks and shoes, insole requirements for patients diagnosed with diabetes mellitus, when to consult a healthcare professional for foot care, and examples of diabetic foot cases with visual examples. Another important aspect of this study is that no study in the literature has been found where preventive diabetic foot education developed in a virtual environment has been implemented using VR headsets. • The training will be provided five times: at baseline, at 4, 8, 12, and 24 weeks. Since patients will be called to the hospital as part of their routine checkups, it will not create any financial or emotional burden.

* The study will include patients who have not previously experienced diabetic foot ulcers. No training program has been found in the literature for patients diagnosed with type 2 diabetes who wear SG glasses. It is believed that this training, unlike traditional learning methods, will provide patients with the opportunity to learn more actively, through hands-on experience, the importance of foot care, how to perform it, and where they have made mistakes in the past.
* This group was chosen because diabetic foot problems are the only complication of diabetes that can be prevented through education. The education provided leads to significant reductions in wound formation and amputations. Preventing diabetic foot problems through education and simple measures is much easier than treating the problem.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with type 2 diabetes at least six months ago
* Those who are over 18 years of age
* Those who volunteer to participate in the study
* Those who can read and write
* Those who have no problems accessing the internet
* Those who have the ability to use a telephone
* Those who do not have sensory losses such as vision or hearing
* Those who do not have communication problems or those who do not have a perception or psychiatric disease diagnosis that would prevent communication
* Those who do not have ulceration in the foot and/or ankle area and/or who have not been diagnosed with diabetic foot will be included in the study.

Exclusion Criteria:

* Individuals who do not meet the criteria for inclusion in the study will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
6 months after giving the first training.The lowest possible score on the Foot Care Behavior Scale (FBS) is 15, and the highest score is 75. A higher scale score indicates that the individual's foot self-care behaviors are better. | Six months
  Diabetic foot training, developed based on literature and expert opinions, will be delivered to patients in the intervention group using virtual reality goggles. The training will cover the importance of diabetes and diabetic foot, risk factors for diabetic foot, causes and symptoms of diabetic foot, preventive foot care practices, how to perform a self-examination of the foot, proper nail care, appropriate sock and shoe selection, insole needs for patients diagnosed with diabetes mellitus, when to consult a healthcare professional for foot care, and examples of diabetic foot cases with visual examples. Patients in the intervention group will receive the diabetic foot training using virtual reality goggles at baseline, 4, 8, 12, and 24 weeks, and will then be administered the Diabetic Foot Behavior Scale. The program will last approximately six months.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep Üniversitesi, Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data of the study will be kept by the researchers.